CLINICAL TRIAL: NCT04479748
Title: DEXTENZA Compared to Topical Steroid Therapy Prior to Cataract Surgery in Patients Who Receive Premium Intraocular Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prism Vision Group (Other)
Responsible Party: Principal Investigator, Dr. Sydney Tyson, Principal Investigator, Prism Vision Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEXTENZA
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Dexamethasone; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextenza insert (Other): Patient's first eye scheduled for surgery will receive an intracanalicular insertion of DEXTENZA (dexamethasone release profile of QID, TID, BID, QD, over 30 days; study eye).
  Interventions: Drug: Dexamethasone
- Fellow-eye (Other): The fellow-eye will receive topical prednisolone acetate 1% (tapering schedule of QID, TID, BID, QD over 30 days). The fellow-eye design in n=30 patients (60 eyes) allows for balance in patient baseline demographic and systemic characteristics.
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: Dexamethasone — Treatment of pain and inflammation following ophthalmic surgery
  Arms: Dextenza insert
Drug: Prednisolone Acetate 1% Oph Susp — Topical steroid
  Arms: Fellow-eye

SUMMARY:
The investigators seek to assess the effect of pre-operative and continued post-operative corticosteroid use on pain, patient preference, visual outcomes, and change in objective quantifiable biological parameters in patients undergoing bilateral cataract surgery with premium intraocular lens implantation with or without baseline ocular surface disease.

Patient's first eye scheduled for surgery will receive an intracanalicular insertion of DEXTENZA (dexamethasone release profile of QID, TID, BID, QD, over 30 days; study eye). The fellow-eye will receive topical prednisolone acetate 1% (tapering schedule of QID, TID, BID, QD over 30 days). The fellow-eye design in n=30 patients (60 eyes) allows for balance in patient baseline demographic and systemic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 or greater with plans to undergo bilateral clear cornea cataract surgery with phacoemulsification and implantation of a premium posterior chamber IOL

  * Schirmer's test score (anesthetized) ≥ 5 mm at Screening in either eye.
  * TBUT ≤ 7 seconds at Screening or Baseline in either eye.
  * All subjects must provide signed written consent prior to participation in any study-related procedures. Able to comply with study requirements and visit schedule.

Exclusion Criteria:

* revious corneal surgery or pathology

  * Active or history of chronic or recurrent inflammatory eye disease in either eye
  * Ocular pain in either eye
  * Proliferative diabetic retinopathy in either eye
  * Significant macular pathology detected on macular optical coherence tomography evaluation at the screening visit in either eye
  * Laser or incisional ocular surgery during the study period and 6 months prior in either eye
  * Prescription and OTC ophthalmic mast cell stabilizers and antihistamines within 21 days prior to Screening and throughout the study period (systemic mast cell stabilizers are allowed, and systemic antihistamines are permitted)
  * Chronic daily use (defined as > 7 consecutive days at the recommended dosing frequency) of systemic narcotics for any chronic pain syndrome (eg, fibromyalgia, rheumatoid arthritis, etc.) during the study period.
  * Ophthalmic artificial tear drop use within 2 hours prior to any study visit. Any OTC artificial tear (preserved or unpreserved) should be continued at the same frequency and with no change in drop brand.
  * Use of any topical prescription ophthalmic medications (including cyclosporine [Restasis®, Cequa®] or topical lifitegrast [Xiidra®], steroids, nonsteroidal anti- inflammatory drugs [NSAIDs], anti-glaucoma medications within 7 days or during study period
  * Participation in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.
  * Corticosteroids (intranasal, inhaled, topical dermatological, and perianal steroids) within 30 days prior to entry in the study are not permitted
  * Pregnant or breast-feeding women, women who wish to become pregnant during the length of study participation, or women of child-bearing potential.
  * Use of systemic NSAID greater than 375 mg per day.
  * Glaucoma or is on medications to treat glaucoma.
  * Ocular Hypertension, defined as IOP of >21 mmHg, is on medications to treat hypertension or has a history of IOP spikes in either eye including steroid-related IOP increases.
  * Presence of nasolacrimal duct obstruction or history of cauterization of the Punctum.
  * Active epiphora or clinically significant dry eye syndrome.
  * Know allergy or sensitivity to the investigational product or its components.
  * The Investigator determines that the subject should not be included for reasons not already specified (e.g, systemic or other ocular disease/abnormality) if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Pain Scale | 30 days
  Proportion of eyes with absence of pain as measured by pain scale (pain score = 0) from Baseline over each time point through Day 30.
  Subjects will use the Ocular Pain Assessment scale. A 0-10 point scale, where 0 is the least pain and 10 is the greatest pain, subjects will be asked to rank their level of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Associates of Vineland, Vineland, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No